CLINICAL TRIAL: NCT01424306
Title: Diet and Systemic Inflammation
Acronym: DASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Mario Kratz, Associate Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NHLBI R21 HL108257; R21HL108257 (NIH)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Low-grade Chronic Inflammation; Intestinal Permeability; Type 2 Diabetes Mellitus; Cardiovascular Disease; Obesity
Keywords: Inflammation; Intestinal permeability; Type 2 diabetes mellitus; Cardiovascular disease; Obesity; Sweetened beverages; Sugar; Fructose; Glucose; High-fructose corn syrup
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fructose-sweetened beverages (Experimental): In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a fructose-sweetened beverage for 8 days.
  Interventions: Other: Fructose-sweetened beverages
- Glucose-sweetened beverages (Experimental): In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a glucose-sweetened beverage for 8 days.
  Interventions: Other: Glucose-sweetened beverages
- High-fructose corn syrup-sweetened beverages (Experimental): In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a high-fructose corn syrup-sweetened beverage for 8 days.
  Interventions: Other: High-fructose corn syrup-sweetened beverages

INTERVENTIONS:
Other: Fructose-sweetened beverages — In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a fructose-sweetened beverage for 8 days. The amount of fructose consumed will be 25% of the subject's estimated daily calorie requirement.
  Arms: Fructose-sweetened beverages
Other: Glucose-sweetened beverages — In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a glucose-sweetened beverage for 8 days. The amount of glucose consumed will be 25% of the subject's estimated daily calorie requirement.
  Arms: Glucose-sweetened beverages
Other: High-fructose corn syrup-sweetened beverages — In addition to consuming a standardized diet, subjects will be asked to consume 4 servings per day of a high-fructose corn syrup-sweetened beverage for 8 days. The amount of high-fructose corn syrup consumed will be 25% of the subject's estimated daily calorie requirement.
  Arms: High-fructose corn syrup-sweetened beverages

SUMMARY:
People with chronic low-grade inflammation have a higher risk for certain diseases such as cardiovascular disease or type 2 diabetes. While it is known that obese people are more likely to show signs of low-grade inflammation than lean individuals, it is unclear what causes this inflammation. In the proposed study, the investigators will examine whether the sugar fructose, when consumed in a sweetened beverage, triggers low-grade inflammation in healthy men and women compared with other caloric sweeteners.

DETAILED DESCRIPTION:
The objective of this proposal is to investigate whether fructose-sweetened beverages trigger low-grade systemic inflammation in healthy men and women. Low-grade systemic inflammation, specifically elevated plasma concentrations of C-reactive protein (CRP), is a risk factor for cardiovascular disease (CVD). While it is known that obesity is associated with inflammation, the causes of low-grade inflammation in humans are not well understood. In a pilot study, the consumption of large amounts of fructose-, but not glucose- or aspartame-sweetened beverages potently induced low-grade inflammation in healthy, lean, young men and women in as little as 8 days. The investigators propose to extend these findings by (a) enrolling a greater number of subjects, (b) enrolling obese as well as non-obese subjects, and (c) including a beverage that is sweetened with high fructose corn syrup (HFCS). HFCS is one of the primary sugars consumed in the United States, and a major source of dietary fructose. Our primary specific aim is to assess whether the consumption of fructose- or HFCS-sweetened beverages promotes systemic low-grade inflammation, as measured by plasma concentrations of CRP and IL-6. The investigators hypothesize that plasma CRP and IL-6 concentrations will be elevated after consumption of fructose-containing beverages (fructose and HFCS) when compared to a glucose-sweetened beverage. Our secondary specific aim is to assess whether the consumption of fructose- or HFCS-sweetened beverages lowers plasma adiponectin concentrations. Specifically, the investigators hypothesize that total and high molecular weight (HMW)-adiponectin concentrations in fasting plasma will be lower after subjects have consumed the fructose- or HFCS-sweetened beverages, compared to a glucose-sweetened beverage.

The investigators will recruit 12 overweight/obese (BMI between 25.0 and 40 kg/m2) and 12 normal weight (BMI between 20 and 24.9 kg/m2) men and women who are free of chronic inflammatory or metabolic disease. In a double-blind, randomized cross-over design, each subject will complete three 8-day standardized dietary periods that will differ only in the type of sweetened beverage administered. Specifically, subjects will be asked to drink four servings of a beverage each day that is sweetened with glucose, fructose, or HFCS (55% fructose, 45% glucose). All solid food will be provided for each of the three 8-day diet periods, and will be consumed ad libitum. Following each dietary period, the investigators will collect fasting blood to measure markers of systemic inflammation and plasma concentrations of total and HMW-adiponectin. We will also assess changes in adipose tissue inflammation and intestinal permeability as potential mechanisms by which fructose-sweetened beverages may trigger systemic inflammation. This study has the potential to identify a dietary trigger of low-grade inflammation, a likely contributor to CVD and metabolic diseases. The public health impact of this project might be considerable given that the consumption of fructose in the population is pervasive, and is modifiable on an individual as well as a population level.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years;
* BMI 20-40 kg/m2;
* Weight stable to within 10 pounds for 6 months prior to entering the study, and at their lifetime maximum weight (or within 30 pounds of it; excluding pregnancy);
* Ability to be admitted for ~30 minutes on three occasions, and ~6 hours on three occasions to the FHCRC Prevention Center;
* Ability to provide informed written consent;
* Willingness to consume only food and beverages provided by the Human Nutrition Laboratory of the FHCRC Prevention Center for three periods of 8 days each.

Exclusion Criteria:

* Presence or history of chronic inflammatory, autoimmune or metabolic diseases;
* Presence of phenylketonuria, hereditary fructose intolerance, fructose malabsorption, or malabsorption syndromes;
* Abuse of alcohol (>2 drinks per day), smoking, or use of recreational drugs;
* Current or recent (within three months) intake of medications likely to interfere with study endpoints (insulin, antidiabetics, β-blockers, anabolic steroids, glucocorticosteroids, daily high-dose non-steroidal anti-inflammatory drugs, warfarin, antibiotics, probiotics);
* Presence of anemia, recent (within 2 months) history of anemia;
* Anyone not willing or able to eat the provided food;
* Current or recent (within 12 months) pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, MS, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] Kuzma JN, Cromer G, Hagman DK, Breymeyer KL, Roth CL, Foster-Schubert KE, Holte SE, Callahan HS, Weigle DS, Kratz M. No difference in ad libitum energy intake in healthy men and women consuming beverages sweetened with fructose, glucose, or high-fructose corn syrup: a randomized trial. Am J Clin Nutr. 2015 Dec;102(6):1373-80. doi: 10.3945/ajcn.115.116368. Epub 2015 Nov 4. PMID 26537945
- [Background] Kuzma JN, Cromer G, Hagman DK, Breymeyer KL, Roth CL, Foster-Schubert KE, Holte SE, Weigle DS, Kratz M. No differential effect of beverages sweetened with fructose, high-fructose corn syrup, or glucose on systemic or adipose tissue inflammation in normal-weight to obese adults: a randomized controlled trial. Am J Clin Nutr. 2016 Aug;104(2):306-14. doi: 10.3945/ajcn.115.129650. Epub 2016 Jun 29. PMID 27357093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 63 volunteers who responded to newspaper advertisements and fliers posted in the Seattle area were screened for eligibility between December 2011 and December 2013.
Pre-assignment Details: Of those 63 volunteers screened, 38 did not meet inclusion criteria and 0 declined to participate. 25 subjects randomized
Groups:
- Fructose - Glucose - HFCS: Subjects treated in the order fructose-sweetened beverage - wash out - glucose-sweetened beverage- wash out - HFCS-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
- Fructose - HFCS - Glucose: Subjects treated in the order fructose-sweetened beverage - wash out - HFCS-sweetened beverage- wash out - glucose-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
- HFCS - Fructose - Glucose: Subjects treated in the order HFCS-sweetened beverage - wash out - fructose-sweetened beverage- wash out - glucose-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
- HFCS - Glucose - Fructose: Subjects treated in the order HFCS-sweetened beverage - wash out - glucose-sweetened beverage- wash out - fructose-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
- Glucose - Fructose - HFCS: Subjects treated in the order glucose-sweetened beverage - wash out - fructose-sweetened beverage- wash out - HFCS-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
- Glucose - HFCS - Fructose: Subjects treated in the order glucose-sweetened beverage - wash out - HFCS-sweetened beverage- wash out - fructose-sweetened beverage
  Treatments each lasted 8 days and were separated by a 20-day washout.
Period: Overall Study
Arm/Group | Fructose - Glucose - HFCS | Fructose - HFCS - Glucose | HFCS - Fructose - Glucose | HFCS - Glucose - Fructose | Glucose - Fructose - HFCS | Glucose - HFCS - Fructose
Started | 4 | 4 | 3 | 3 | 5 | 6
Completed | 4 | 4 | 3 | 3 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only results of 24 subjects who completed study 'per protocol' are reported here
Groups:
- Study Subjects: All six treatment orders combined
Arm/Group | Study Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (4.8)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 92 (10)
Physical activity [Mean (Standard Deviation); unit: MET-hr/wk] | 68.7 (45.9)
Estimated total calorie requirement [Mean (Standard Deviation); unit: kcal/d] | 2560 (370)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Plasma C-reactive Protein
Description: The concentration of C-reactive protein in fasting plasma will be measured by high-sensitivity assay at the beginning (day 1) and end (day 9) of each 8-day dietary period.
Time Frame: Beginning (day 1) and end (day 9) of each diet period.
Population: All completed participants combined in per protocol analysis
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Fructose Arm - Day 1: CRP measured on day 1 of fructose-sweetened beverage intervention period
- Fructose Arm - Day 9: CRP measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 1: CRP measured on day 1 of glucose-sweetened beverage intervention period
- Glucose Arm - Day 9: CRP measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 1: CRP measured on day 1 of HFCS-sweetened beverage intervention period
- HFCS Arm - Day 9: CRP measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 1 | Fructose Arm - Day 9 | Glucose Arm - Day 1 | Glucose Arm - Day 9 | HFCS Arm - Day 1 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
mg/L | 0.91 [0.45 to 2.35] | 1.07 [0.48 to 2.10] | 1.67 [0.36 to 2.91] | 1.09 [0.38 to 3.04] | 1.18 [0.38 to 2.49] | 0.84 [0.49 to 2.48]
Statistical Analysis 1: Comparison: Fructose Arm - Day 1 vs Fructose Arm - Day 9 vs Glucose Arm - Day 1 vs Glucose Arm - Day 9 vs HFCS Arm - Day 1 vs HFCS Arm - Day 9; RM-ANOVA; Test type: Other; p = 0.403, RM-ANOVA — P value for the time x diet interaction reflects overall comparison of 3 dietary phases by RM-ANOVA

2. Primary Outcome: Fasting Plasma Interleukin-6 on Day 9 of Each Diet Period
Description: The concentration of interleukin-6 in fasting plasma will be measured by high-sensitivity enzyme-linked immunosorbent assay at the end (day 9) of each 8-day dietary period.
Time Frame: End (day 9) of each diet period
Population: All completed participants combined in per protocol analysis
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Fructose Arm - Day 9: IL-6 measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: IL-6 measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: IL-6 measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24
pg/mL | 0.97 [0.62 to 1.90] | 1.14 [0.61 to 1.95] | 0.96 [0.61 to 1.79]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.933, RM-ANOVA — P-diet: reflects an overall comparison of the 3 dietary phases by RM-ANOVA

3. Secondary Outcome: Fasting Plasma Adiponectin
Description: The concentration of adiponectin in fasting plasma will be measured by enzyme-linked immunosorbent assay at the end (day 9) of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: All completed participants combined in per protocol analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fructose Arm - Day 9: Adiponectin measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: Adiponectin measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: Adiponectin measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 4635 (2545) | 4353 (2198) | 4514 (2195)
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.196, RM-ANOVA — P-diet: reflects an overall comparison of the 3 dietary phases by RM-ANOVA

4. Secondary Outcome: Mean Daily Calorie Intake
Description: Mean daily calorie intake will be assessed during each of the three 8-day diet periods. All foods will be provided to the subjects in excess of what they are estimated to require, and calorie intake will be assessed by subtracting returned foods from foods administered.
Time Frame: The mean daily calorie intake during each of the 8-day diet periods will be calculated.
Population: All completed participants combined in per protocol analysis
Measure: Mean (Standard Deviation); unit: kcal/d
Groups:
- Fructose Arm: Average total energy consumed each day during the fructose-sweetened beverage intervention period
- Glucose Arm: Average total energy consumed each day during the glucose-sweetened beverage intervention period
- HFCS Arm: Average total energy consumed each day during the HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm | Glucose Arm | HFCS Arm
Number analyzed (Participants) | 24 | 24 | 24
kcal/d | 2970 (482) | 2940 (460) | 2950 (535)
Statistical Analysis 1: Comparison: Fructose Arm vs Glucose Arm vs HFCS Arm; Test type: Other — RM-ANOVA; p = 0.880, RM-ANOVA — Reflects an overall comparison of the 3 dietary phases by RM-ANOVA

5. Secondary Outcome: Intestinal Permeability, as Assessed by the 5-hour Urinary Lactulose/Mannitol Test
Description: Intestinal permeability will be assessed on day 9 of each diet period by administering a beverage containing 2 g of mannitol and 5 g of lactulose followed by collecting urine for 5 hours afterwards. Recovery of mannitol and lactulose in urine will be measured by gas chromatography, and will be indicative of the degree of intestinal permeability.
Time Frame: End (day 9) of each diet period.
Population: All completed participants combined in per protocol analysis
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Fructose Arm - Day 9: Lactulose:Mannitol ratio measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: Lactulose:Mannitol ratio measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: Lactulose:Mannitol ratio measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24
ratio | 0.047 [0.031 to 0.054] | 0.043 [0.031 to .048] | 0.031 [0.026 to 0.035]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p < 0.001, Repeated measures ANOVA — P-value reflects an overall comparison of the 3 dietary phases by RM-ANOVA

6. Secondary Outcome: Fasting Plasma Zonulin Concentrations
Description: Zonulin concentrations will be measured by enzyme-linked immunosorbent assay in fasting plasma collected on day 9 of each diet period. Plasma zonulin is a marker of intestinal permeability.
Time Frame: End (day 9) of each diet period.
Population: All completed participants combined in per protocol analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fructose Arm - Day 9: Zonulin measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: Zonulin measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: Zonulin measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 12.78 (1.54) | 12.69 (1.70) | 12.92 (1.49)
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.366, RM-ANOVA — P-value reflects an overall comparison of the 3 dietary phases by RM-ANOVA

7. Secondary Outcome: Fasting Plasma Lipopolysaccharide-binding Protein (LBP)
Description: Lipopolysaccharide-binding protein (LBP) will be measured by enzyme-linked immunosorbent assay in fasting plasma collected on day 9 of each diet period. LBP is an acute phase protein secreted by the liver in response to endotoxin (lipopolysaccharide) exposure.
Time Frame: End (day 9) of each diet period.
Population: All completed participants combined for protocol analysis
Measure: Median (Inter-Quartile Range); unit: ug/mL
Groups:
- Fructose Arm - Day 9: LBP measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: LBP measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: LBP measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 24 | 24 | 24
ug/mL | 27.7 [19.8 to 34.2] | 26.1 [21.7 to 40.0] | 29.8 [21.5 to 36.0]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.387, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

8. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of TNF-alpha mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of TNF-alpha mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Mean (Standard Deviation); unit: copy number/ng total RNA
Groups:
- Fructose Arm - Day 9: Gene expression measured on day 9 of fructose-sweetened beverage intervention period
- Glucose Arm - Day 9: Gene expression measured on day 9 of glucose-sweetened beverage intervention period
- HFCS Arm - Day 9: Gene expression measured on day 9 of HFCS-sweetened beverage intervention period
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 1.40 (0.58) | 1.44 (0.89) | 1.24 (0.67)
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.476, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

9. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of IL-1beta mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of IL-1beta mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Median (Inter-Quartile Range); unit: copy number/ng total RNA
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 0.41 [0.26 to 0.54] | 0.33 [0.25 to 0.41] | 0.32 [0.27 to 0.84]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.596, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

10. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of IL-6 mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of IL-6 mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Median (Inter-Quartile Range); unit: copy number/ng total RNA
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 0.53 [0.35 to 0.74] | 0.49 [0.37 to 0.58] | 0.51 [0.38 to 0.75]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.492, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

11. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of IL-10 mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of IL-10 mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Median (Inter-Quartile Range); unit: copy number/ng total RNA
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 0.66 [0.34 to 1.14] | 0.90 [0.65 to 1.19] | 0.95 [0.34 to 1.44]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.149, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

12. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of CCL2 mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of CCL2 mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Median (Inter-Quartile Range); unit: copy number/ng total RNA
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 31.5 [22.9 to 47.6] | 27.2 [22.6 to 33.6] | 25.3 [19.3 to 34.4]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.056, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

13. Secondary Outcome: Adipose Tissue Inflammation - Tissue Expression of IFN-gamma mRNA
Description: A subgroup of the study population will be enrolled into an ancillary study that will aim to assess the effects of consuming fructose- vs. high-fructose corn syrup- vs. glucose-sweetened beverages on adipose tissue inflammation. Adipose tissue inflammation will be assessed by whole adipose tissue gene expression analysis of IFN-gamma mRNA. Abdominal subcutaneous adipose tissue samples will be obtained from subjects enrolled into the ancillary study by needle aspiration biopsy on day 9 of each 8-day dietary period.
Time Frame: End (day 9) of each diet period.
Population: A subset of the study population opted to undergo voluntary adipose tissue biopsy
Measure: Median (Inter-Quartile Range); unit: copy number/ng total RNA
Arm/Group | Fructose Arm - Day 9 | Glucose Arm - Day 9 | HFCS Arm - Day 9
Number analyzed (Participants) | 14 | 14 | 14
copy number/ng total RNA | 0.23 [0.15 to 0.44] | 0.20 [0.15 to 0.27] | 0.23 [0.17 to 0.38]
Statistical Analysis 1: Comparison: Fructose Arm - Day 9 vs Glucose Arm - Day 9 vs HFCS Arm - Day 9; Test type: Other — RM-ANOVA; p = 0.520, RM-ANOVA — P-value reflects overall comparison of the 3 dietary phases by RM-ANOVA

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 years.
Groups:
- Fructose Arm: Powdered fructose mixed with powdered drink flavoring (Lemon)
- Glucose Arm: Powdered dextrose mixed with powdered drink flavoring (Lemon) and aspartame to match sweetness
- HFCS Arm: HFCS liquid mixed with powdered drink flavoring (Lemon) and aspartame to match sweetness
Arm/Group | Fructose Arm | Glucose Arm | HFCS Arm
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 1/25 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fructose Arm (N=24) | Glucose Arm (N=25) | HFCS Arm (N=24)
Bruise from abdominal needle aspiration biospy (Skin and subcutaneous tissue disorders) | 1/14 (1) | 1/14 (1) | 0/13 (0)
Gastrointestinal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Gastrointestinal discomfort including cramping, bloating, and/or diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No